CLINICAL TRIAL: NCT02074774
Title: Comparison of the IntellO2 - Precision Flow Automatic FiO2 Controller to Manual Control for Optimizing Oxygenation in Preterm Infants Receiving High Flow Nasal Cannula Therapy
Brief Title: IntellO2 vs Manual Control for Optimizing Oxygenation in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vapotherm, Inc. (Industry)
Collaborators: Ashford and St. Peter's Hospitals NHS Trust (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RP-NIAE2014001Reg
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Oxygen Titration in Preterm Infants to Manage Lung Disease
Keywords: nasal cannula, high flow oxygen therapy, pulse oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IntellO2 (Experimental): Automated control of FiO2
  Interventions: Device: IntellO2
- Manual (Active Comparator): Manual control of FiO2
  Interventions: Other: Manual control

INTERVENTIONS:
Device: IntellO2 — Automated FiO2 regulator that responds to pulse oximetry measures
  Arms: IntellO2
Other: Manual control — Standard practice of manually titrating FiO2 as needed.
  Arms: Manual

SUMMARY:
The overall objective of this study is to demonstrate that the IntellO2 device providing automated control of fraction of inspired oxygen (FiO2) adjustments in spontaneously breathing infants with fluctuating arterial blood oxygen saturation levels is safe and efficacious in the routine clinical environment. Specifically, it is hypothesized that the IntellO2 will perform as well or better than standard practice for maintaining infants' arterial blood oxygen saturation in a target range while minimizing the exposure to elevated levels of oxygen in the inspired gas.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants being treated with high flow nasal cannula therapy
2. A need for supplemental oxygen as demonstrated by an required FiO2 > 0.25 at enrollment
3. Requiring a flow rate of greater than 2 L/min such that the assumed inspired oxygen fraction matched delivered oxygen fraction (definition of HFNC).

Exclusion Criteria:

1. Major congenital abnormalities
2. Hemodynamic instability, defined as being outside of a normotensive range based on each infant's individual characteristics
3. Seizures
4. Ongoing sepsis
5. Meningitis
6. Clinician's concern regarding stability of the infant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Percent time in target range for oxygen saturation by pulse oximetry | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reynolds, MB.BS PhD, Principal Investigator — Ashford and St. Peter's Hospitals NHS Trust; George C Dungan, MPhil, Study Director — Vapotherm, Inc.
Locations (2):
- United Kingdom (2):
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - Ashford and St. Peter's Hospitals NHS Trust, Chertsey, Surrey

REFERENCES:
- [Derived] Reynolds PR, Miller TL, Volakis LI, Holland N, Dungan GC, Roehr CC, Ives K. Randomised cross-over study of automated oxygen control for preterm infants receiving nasal high flow. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F366-F371. doi: 10.1136/archdischild-2018-315342. Epub 2018 Nov 21. PMID 30464005